CLINICAL TRIAL: NCT01761162
Title: ProMRI Study of the Entovis Pacemaker System
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: G120226
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Safety of the ProMRI Pacemaker System Under Specific MRI Conditions
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker Therapy: Patients with a ProMRI Pacemaker System
  Interventions: Device: Patients with a ProMRI Pacemaker System; Other: Magnetic Resonance Imaging (MRI) scan

INTERVENTIONS:
Device: Patients with a ProMRI Pacemaker System — Bradycardia Slow Heart Beat
Other: Magnetic Resonance Imaging (MRI) scan — MRI scan of head and lower back.

SUMMARY:
The objective of the ProMRI Study is to demonstrate the clinical safety of the ProMRI Pacemaker System when used under specific MRI conditions.

ELIGIBILITY:
Inclusion Criteria:

The following initial inclusion criteria must be met for a subject to be enrolled and considered for the MRI-procedure:

* Age greater than 18 years
* Subject body height greater than 140 cm (4' 7")
* Able and willing to complete MRI testing
* Able to provide written informed consent
* Available for follow-up visit at the study site
* Implanted with a pacemaker system consisting only of an Entovis pacemaker (DR-T, SR-T) and one or two Setrox S 53 or Setrox S 60 pacemaker lead(s). (No leads other than Setrox S (53 or 60 cm) leads may be implanted. This includes lead extensions or abandoned leads in the subject.)
* Pacemaker implanted pectorally
* All pacemaker system components implanted, repositioned, or exchanged at least 5 weeks prior to enrollment
* Underling rhythm identifiable during sensing test
* All pacing thresholds are measureable and are less than or equal to 2.0 V @0.4 ms
* Absence of phrenic nerve stimulation at 4.8V @ 1.0 ms
* Pacing impedance is between 200 and 1500 ohm
* Able and willing to use the Cardio Messenger

At the pre-MRI procedure, the following procedure-related criteria must be met for the subject to undergo the MRI scan:

* Absence of phrenic nerve stimulation at 4.8V @ 1.0 ms
* |pacing threshold at Pre-MRI follow-up - pacing threshold at baseline| ≤ 0.5 V
* All pacing thresholds are measureable and are ≤ 2.0 V @ 0.4 ms
* The pacemaker system has been implanted for at least 6 weeks.
* Subject did not have a pacemaker or lead explant, exchange or reposition in the previous 6 weeks.
* All lead impedances are between 200 and 1500 ohm.
* Battery status is at least 30% of capacity

Exclusion Criteria:

* Enrolled in any other clinical study
* For pacemaker systems that include an atrial lead, subjects with either

  * Persistent atrial arrhythmia (lasting longer than 7 days or requiring cardioversion)
  * Permanent atrial arrhythmia
* Life expectancy of less than three months
* Pregnancy
* Cardiac surgery expected in the next three months
* Implanted with other medical devices that may interact with MRI, such as:

  * abandoned pacemaker/ICD leads
  * lead extensions
  * mechanical valves
  * other active medical devices
  * non-MRI compatible devices
  * other metallic artifacts/components in body that may interact with MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigators' general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - John Muir Medical Center, Concord, California
  - Hoag Hospital, Newport Beach, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Valparaiso, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Louisiana Heart Rhythm Specialists, Lafayette, Louisiana
  - Cumberland, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Burlington, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Joseph Mercy Medical Center, Ypsilanti, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Camden, New Jersey
  - New York Hospital Queens, Flushing, New York
  - New York, New York
  - Winston-Salem, North Carolina
  - Toledo Hospital, Toledo, Ohio
  - Saint Mary Medical Center, Langhorne, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Greenville, South Carolina
  - Richmond, Virginia

REFERENCES:
- [Result] Bailey WM, Rosenthal L, Fananapazir L, Gleva M, Mazur A, Rinaldi CA, Kypta A, Merkely B, Woodard PK; ProMRI/ProMRI AFFIRM Study Investigators. Clinical safety of the ProMRI pacemaker system in patients subjected to head and lower lumbar 1.5-T magnetic resonance imaging scanning conditions. Heart Rhythm. 2015 Jun;12(6):1183-91. doi: 10.1016/j.hrthm.2015.02.010. Epub 2015 Feb 11. PMID 25680307

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pacemaker Therapy
Started | 229
Completed | 226
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (10.7)
Gender [Count of Participants; unit: Participants]
  Female | 71
  Male | 158

OUTCOME MEASURES:

1. Primary Outcome: MRI and Pacing System Related Serious Adverse Device Effect (SADE) Free Rate
Time Frame: 1 Month Post-MRI
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 229
percentage of participants | 100 [98.4 to 100]

2. Primary Outcome: Percentage of Participants Free of Atrial Pacing Threshold Rise
Description: Evaluate the percentage of atrial pacing leads free of pacing threshold increase between the pre-MRI and one-month post-MRI follow-up.
Time Frame: Pre-MRI, 1 Month Post-MRI
Population: Number of participants with an atrial lead and same atrial threshold polarity (either uni- or bipolar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 191
percentage of participants | 99.0 [96.3 to 99.9]

3. Primary Outcome: Percentage of Participants Free of Ventricular Pacing Threshold Rise
Description: Evaluate the percentage of ventricular pacing leads free of pacing threshold increase between the Pre-MRI and one-month post-MRI follow-up.
Time Frame: Pre-MRI, 1 Month Post-MRI
Population: Number of participants with a ventricular lead and same ventricular threshold polarity (either uni- or bipolar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 217
percentage of participants | 100 [98.3 to 100]

4. Primary Outcome: Percentage of Participants Free of P-wave Sensing Attenuation
Description: Evaluate the percentage of subjects free of P-wave attenuation between the pre-MRI and one-month post-MRI follow-up.
Time Frame: Pre-MRI, 1 Month Post-MRI
Population: Number of participants with an atrial lead and same atrial sensing polarity (either uni- or bipolar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 168
percentage of participants | 99.4 [96.7 to 100]

5. Primary Outcome: Percentage of Participants Free of R-wave Sensing Attenuation
Description: Evaluate the percentage of subjects free of R-wave attenuation between the pre-MRI and one-month post-MRI follow-up.
Time Frame: Pre-MRI, 1 Month Post-MRI
Population: Number of participants with a ventricular lead and same ventricular sensing polarity (either uni- or bipolar) at pre-MRI and one-month post-MRI.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pacemaker Therapy
Number analyzed (Participants) | 194
percentage of participants | 99.5 [97.2 to 100]

ADVERSE EVENTS:
Arm/Group | Pacemaker Therapy
Serious Adverse Events (participants affected / at risk) | 21/229
Other Adverse Events (participants affected / at risk) | 30/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker Therapy (N=229)
Angina (Cardiac disorders) | 2 (2)
Arrhythmia (Cardiac disorders) | 2 (2)
Arterial Stenosis (Vascular disorders) | 2 (2)
Coronary Artery Disease (Vascular disorders) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Myocardial Infarction (Vascular disorders) | 1 (1)
Mild to moderate post-operative risks (General disorders) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (3)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Syncope/Pre-Syncope (Vascular disorders) | 3 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker Therapy (N=229)
Arrythmia (Cardiac disorders) | 13 (14)
MRI Incidental Finding (General disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators agree to submit copies of any manuscript proposed for publication to Sponsor for review at least 30 days in advance of submission for publication or presentation. Sponsor may extend such review period for another 90 days to file patent applications or take other steps to protect its intellectual property interests, or to remove from the paper or presentation any language that is detrimental to Sponsor's intellectual property interests.